CLINICAL TRIAL: NCT02985216
Title: A Randomized, Double-blind, Active-Controlled, Multi-center, Phase 3 Trial to Compare the Safety and Efficacy Between YHD1119 and Pregabalin in Patients With Peripheral Neuropathic Pain
Brief Title: Clinical Trial of YHD1119 in Patients With Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YHD1119-301
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2017-02

CONDITIONS: Peripheral Neuropathic Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YHD1119 (Experimental): YHD1119 150mg for the first 1 week, then forced titrated to YHD1119 300mg for the 1 week. And then YHD1119 150~600mg for the 2 weeks, then YHD1119 fixed dose was administrated for 8 weeks.
  Interventions: Drug: YHD1119
- Lyrica (Active Comparator): Lyrica 150mg for the first 1 week, then forced titrated to Lyrica 300mg for the 1 week. And then Lyrica 150~600mg for the 2 weeks, then Lyrica fixed dose was administrated for 8 weeks.
  Interventions: Drug: Lyrica

INTERVENTIONS:
Drug: YHD1119 — YHD1119 150mg, PO YHD1119 300mg, PO
  YHD1119 600mg, PO
  Other Names: Pregabalin
  Arms: YHD1119
Drug: Lyrica — Lyrica 75mg, PO Lyrica 150mg, PO Lyrica 300mg, PO
  Other Names: Pregabalin
  Arms: Lyrica

SUMMARY:
A Randomized, Double-blind, Active-Controlled, Multi-center, Phase 3 Trial to Compare the Safety and Efficacy between YHD1119 and Pregabalin in Patients with Peripheral Neuropathic Pain

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* HbA1c ≤ 9.5% diabetes mellitus patients with pain over 6 months in Diabetic Peripheral Neuropathy or postherpetic Neuralgia patients at least 3 months pain after diagnosis of skin rash due to herpes zooster

Exclusion Criteria:

* Have Brittle diabetes mellitus

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Change From Baseline to End of Treatment (EOT) in Weekly Mean Pain Score on the Daily Pain Rating Scale (DPRS) | Baseline, Day 85

SECONDARY OUTCOMES:
Change From Baseline in Mean Pain Score on the Daily Pain Rating Scale (DPRS) | Day 1, 8, 15, 22, 29, 57, 85
Mean Pain Score on the Daily Pain Rating Scale at each visit | Day 1, 8, 15, 22, 29, 57, 85
Patients proportion of reduction over 30% in Mean Pain Score from Baseline | Day 1, 8, 15, 22, 29, 57, 85
Change of duration-modification from baseline in Mean Pain Score on the Daily Pain Rating Scale (DPRS) | Day 1, 8, 15, 22, 29, 57, 85
Patient Global Impression of Change (PGIC) | Day 85
Clinical Global Impression of Change (CGIC) | Day 85
SF-12 (Short form-12) | Baseline, Day 85
C-SSRS (Columbia Suicide Severity Rating Scale) | Baseline, Day 8, 29, 85

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chul KIM, M.D.,Ph.D., Principal Investigator — Seoul National University
Locations (1):
- Yong Chul Kim, Seoul, South Korea